CLINICAL TRIAL: NCT03077360
Title: Skeletal Muscle Diacylglycerol and Sphingolipids - Impact of Localization and Species on Insulin Resistance in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16-1404; 5R01DK111559 (NIH)
Record Dates: First submitted 2017-03-01; First posted 2017-03-10 (Actual); Results first posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Mellitus, Type 2; Pre-diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Weight loss only (Experimental)
  Interventions: Behavioral: Lifestyle
- Exercise Only (Experimental)
  Interventions: Behavioral: Lifestyle
- Delayed Intervention Control (No Intervention)

INTERVENTIONS:
Behavioral: Lifestyle — Lifestyle changes to lose weight or become more fit
  Arms: Exercise Only; Weight loss only

SUMMARY:
The rationale for the proposed research is that elucidating changes in localized diacylglycerol (DAG) and sphingolipid species that predict insulin sensitivity will reveal specific localized lipids to target in therapeutics for type 2 diabetes. To attain the overall objective, the investigators propose three specific aims: 1. Identify the influence of sarcolemmal DAG and sphingolipids on cell signaling and insulin sensitivity before and after insulin sensitizing lifestyle interventions. Strong preliminary data shape the hypothesis that sarcolemmal 1,2-disaturated DAG and C18:0 ceramide species will decrease after insulin sensitizing lifestyle interventions, leading to less Protein kinase C (PKC) and Protein phosphatase 2A (PP2A) activation, and enhanced insulin signaling. Skeletal muscle DAG and sphingolipid isomers, species, localization, and de novo synthesis will be measured before and after diet-induced weight loss or exercise training interventions in obese men and women. Insulin sensitivity will be measured using insulin clamps, and muscle lipids using Liquid Chromatography Mass Spectrometry (LC/MS). 2. Determine the impact of mitochondrial/ER (endoplasmic reticulum) DAG and sphingolipids on mitochondrial function and ER stress in vivo, before and after insulin sensitizing lifestyle interventions. The investigators hypothesize, again based on preliminary data, that mitochondrial/ER sphingolipids will decrease, yet DAG will increase after insulin sensitizing lifestyle interventions, and each will associate with increased insulin sensitivity. Changes in sphingolipids will relate to increased mitochondrial function, less ER stress, reactive oxygen species (ROS), and acyl-carnitine formation, while changes in DAG will relate to increased mitochondrial content and dynamics. 3. Identify the effect of exogenous DAG and sphingolipids on mitochondrial function in vitro, before and after insulin sensitizing lifestyle interventions. The working hypothesis is that DAG and sphingolipids will reduce mitochondrial respiration and increase ROS and acyl-carnitine content, but will be attenuated after endurance exercise training. The proposed research is innovative because it represents a substantive departure from the status quo by addressing cellular compartmentalization of bioactive lipids. The investigators contribution will be significant by identifying key species and locations of DAG and sphingolipids promoting insulin resistance, as well as mechanisms explaining accumulation that could be modified by insulin sensitizing therapeutic interventions.

DETAILED DESCRIPTION:
Accumulation of bioactive lipids such as diacylglycerol (DAG) and sphingolipids are one mechanism proposed to promote muscle insulin resistance. Recent data indicate these lipids are located in membranes, but the distribution and signaling of DAG and sphingolipids in specific cellular organelles which regulate insulin sensitivity is not known. There is a critical need to address these gaps in knowledge to design appropriate interventions to prevent and treat lipid-induced insulin resistance. The overall objective of this project is to determine the impact of changes in subcellular DAG and sphingolipid species, signaling, and metabolic function before and after insulin sensitizing lifestyle interventions. The investigators central hypothesis is that DAG and sphingolipids in muscle promote insulin resistance via mechanisms that are unique to location, type of lipid, and species. The rationale for the proposed research is that elucidating changes in localized DAG and sphingolipid species that predict insulin sensitivity will reveal specific localized lipids to target in therapeutics for type 2 diabetes. To attain the overall objective, the investigators propose three specific aims: 1. Identify the influence of sarcolemmal DAG and sphingolipids on cell signaling and insulin sensitivity before and after insulin sensitizing lifestyle interventions. Strong preliminary data shape the hypothesis that sarcolemmal 1,2-disaturated DAG and C18:0 ceramide species will decrease after insulin sensitizing lifestyle interventions, leading to less Protein kinase C (PKC) and Protein phosphatase 2A (PP2A) activation, and enhanced insulin signaling. Skeletal muscle DAG and sphingolipid isomers, species, localization, and de novo synthesis will be measured before and after diet-induced weight loss or exercise training interventions in obese men and women. Insulin sensitivity will be measured using insulin clamps, and muscle lipids using Liquid Chromatography Mass Spectrometry (LC/MS). 2. Determine the impact of mitochondrial/ER (endoplasmic reticulum) DAG and sphingolipids on mitochondrial function and ER stress in vivo, before and after insulin sensitizing lifestyle interventions. The investigators hypothesize, again based on preliminary data, that mitochondrial/ER sphingolipids will decrease, yet DAG will increase after insulin sensitizing lifestyle interventions, and each will associate with increased insulin sensitivity. Changes in sphingolipids will relate to increased mitochondrial function, less ER stress, reactive oxygen species (ROS), and acyl-carnitine formation, while changes in DAG will relate to increased mitochondrial content and dynamics. 3. Identify the effect of exogenous DAG and sphingolipids on mitochondrial function in vitro, before and after insulin sensitizing lifestyle interventions. The working hypothesis is that DAG and sphingolipids will reduce mitochondrial respiration and increase ROS and acyl-carnitine content, but will be attenuated after endurance exercise training. The proposed research is innovative because it represents a substantive departure from the status quo by addressing cellular compartmentalization of bioactive lipids. The investigators contribution will be significant by identifying key species and locations of DAG and sphingolipids promoting insulin resistance, as well as mechanisms explaining accumulation that could be modified by insulin sensitizing therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 30-40 kg/m2
* Planned physical activity: <2 hrs/week
* Glucose tolerance:

  1. Normal glucose tolerance (NGT) defined as:

     1. HbA1c of <5.7%,
     2. pre-diabetes as HbA1c of 5.7-6.4%, and
     3. type 2 diabetes as HbA1c of ≥6.5%
  2. pre-diabetes, and
  3. Type 2 diabetes
* Oral contraceptive use: Yes or No as long as there is no change during the study
* Thyroid status: TSH between 0.5-5.0 mU/L

Exclusion Criteria:

* Currently taking

  1. Thiazolidinediones
  2. Insulin
* Pregnant
* Smoker (tobacco and any form of marijuana use)
* Fasting triglycerides >400mg/dl

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2020-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Bergman, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 14 participants dropped out of the study prior to randomization.
Groups:
- Delayed Intervention Control: Control group, no intervention. Participants were offered all benefits of the interventions after study completion.
Period: Overall Study
Arm/Group | Weight Loss Only | Exercise Only | Delayed Intervention Control
Started | 17 | 17 | 14
Completed | 17 | 16 | 12
Not Completed | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Demographics data was only collected for participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Weight Loss Only | Exercise Only | Delayed Intervention Control | Total
Number analyzed (Participants) | 17 | 16 | 12 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (2.4) | 39.6 (3.1) | 39.8 (2.7) | 39.65 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 6 | 23
  Male | 8 | 8 | 6 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 5
  Not Hispanic or Latino | 16 | 14 | 10 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 5
  White | 15 | 13 | 9 | 37
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 12 | 45

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Insulin Sensitivity Compared to Baseline Measurement.
Description: Hyperinsulinemic/euglycemic clamp measured as glucose infusion rate in mg/kg/min.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Weight Loss Only | Exercise Only | Delayed Intervention Control
Number analyzed (Participants) | 17 | 16 | 12
Percent change | 31.8 (8.8) | 17.4 (8.7) | -4.8 (9.3)

2. Primary Outcome: Percent Change in Localized Muscle Lipids Compared to Baseline
Description: We measured changes in sarcolemmal, mitochondrial, nuclear and cytosolic lipids measured in pmol/ug protein after compared to before the interventions
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: percentage change
Groups:
- Delayed Intervention Control: Free living control group which performed intervention of their choice after finishing
Arm/Group | Weight Loss Only | Exercise Only | Delayed Intervention Control
Number analyzed (Participants) | 18 | 16 | 12
percentage change
  Mitochondrial triglyceride | -25 (6) | -30 (7) | 5 (6)
  Nuclear triglyceride | -20 (5) | -25 (5) | 10 (3)
  Nuclear 1,2-Diacylglycerol | 20 (4) | 25 (5) | -5 (1)

3. Primary Outcome: Percent Change in Body Weight Compared to Baseline Measurement
Description: This is the percent change in body weight for each group after the 12 week intervention.
Time Frame: Baseline, 3 Months
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Weight Loss Only | Exercise Only | Delayed Intervention Control
Number analyzed (Participants) | 17 | 16 | 12
Percent | -10.5 (0.9) | -0.5 (0.5) | 0.5 (0.4)

ADVERSE EVENTS:
Time Frame: 3 Months
Arm/Group | Weight Loss Only | Exercise Only | Delayed Intervention Control
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16 | 0/12
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/60/NCT03077360/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT03077360/ICF_001.pdf